CLINICAL TRIAL: NCT00035672
Title: Genetic Predictors of Incident Cardiovascular Disease
Status: Withdrawn | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sharon L.R. Kardia, Professor of Epidemiology, University of Michigan
Other Study IDs: 997; R01HL068737 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
To evaluate how current genetic information about cardiovascular disease susceptibility genes contributes to the prediction of future cardiovascular disease outcomes.

DETAILED DESCRIPTION:
BACKGROUND:

During the 1980s and 1990s, genetic research in cardiovascular disease (CVD), as well as other common chronic diseases, has been dominated by single gene linkage and association studies focused on understanding of the genetics of prevalent disease. Rarely have there been studies of the longitudinal predictive value of these genetic variations. Furthermore, few studies have attempted to address the complex and high-dimensional genetic reality that underlies an individual's risk of disease. A crucial next step in CVD genetic research is the evaluation of the contribution of variations in many genes simultaneously, and their interactions with traditional risk factors, to the longitudinal prediction of CVD in individuals and families.

DESIGN NARRATIVE:

The study uses participants from the Rochester Family Heart Study (RFHS) which provides one of the richest genetic epidemiological resources for this type of study. The RFHS represents 3941 individuals distributed among 552 three- generation pedigrees ascertained without regard to health status during two phases of collection. Phase I was from 1984 - 1988 and Phase II was from 1988 - 1991. These participants have extensive demographic, physiological, genetic, and clinical information measured at baseline. This study builds upon this already established resource by conducting a longitudinal follow-up of the RFHS participants to address two central questions: 1) Do measured genetic variations in known susceptibility genes provide additional predictive information about risk of future CVD outcomes beyond the information provided by more traditional risk factors? and 2) Do these measured genetic variations explain patterns of disease aggregation in families and can these patterns be used to predict disease in future generations?

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Kardia — University of Michigan

REFERENCES:
- [Background] Kardia SL, Modell SM, Peyser PA. Family-centered approaches to understanding and preventing coronary heart disease. Am J Prev Med. 2003 Feb;24(2):143-51. doi: 10.1016/s0749-3797(02)00587-1. PMID 12568820
- [Background] Sing CF, Stengard JH, Kardia SL. Dynamic relationships between the genome and exposures to environments as causes of common human diseases. World Rev Nutr Diet. 2004;93:77-91. doi: 10.1159/000081252. No abstract available. PMID 15496802